CLINICAL TRIAL: NCT01493648
Title: Muscle-Related Side Effects of Statins: Functional Impact, Mechanisms, and Potential Relief With Vitamin D Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: MOP 114917
Record Dates: First submitted 2011-11-29; First posted 2011-12-16 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: HMG COA Reductase Inhibitor Adverse Reaction
Keywords: statins; side effects; muscle; vitamin D; biopsy; strength; fatigue
MeSH Terms: conditions — Fatigue | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental)
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — Participants will receive weekly doses of 30,000 IU of vitamin D for 3 months.
  Other Names: Cholecalciferol, D-tabs
  Arms: Vitamin D
Drug: Placebo — Participants will receive placebo (lactose 100 mg) for 3 months.
  Arms: Placebo

SUMMARY:
This proposal will explore muscle function (strength and endurance) in men and women suffering from statin-induced muscle symptoms. The mechanisms responsible for these muscle symptoms will be explored. Also, the investigators will assess the potential usefulness of vitamin D supplementation in a randomized control trial.

DETAILED DESCRIPTION:
Statins are a class of drugs that are widely prescribed to lower blood cholesterol levels. Although they have few side effects, many patients report muscle pain, cramps, and weakness when using these drugs. We know very little on the real impact of these muscle symptoms on patient quality of life, especially in relation to muscle strength and endurance.

Patients under statin therapy will stop medication for 2 months. Results from blood sample, muscle function and muscle biopsy (in some participants) will be compared with baseline. Participants will then take vitamin D supplementation or placebo for one month. Thereafter, statin will be reintroduced for two months while continuing vitamin D or placebo supplementation. At the end of that time, measures from blood sample, muscle function and muscle biopsy will be compared with other visits.

ELIGIBILITY:
Inclusion Criteria:

* statin therapy
* healthy and sedentary or moderately physical active

Exclusion Criteria:

* Current treatment with other lipid-lowering drugs
* Natural medicine affecting lipid metabolism
* CK levels above the normal range
* Clinical vitamin D deficiency
* Impaired liver or kidney function
* Untreated hypo- or hyperthyroidism
* Treatment with other medications known to increase risk of myopathy
* Existing infection requiring antibiotic therapy
* Consumption of greater than 60 ml of grapefruit juice per day
* Inherited muscle disorders or myopathy
* Polymyositis or inflammatory myopathy
* Use of corticosteroids
* Comorbidities resulting in muscle or bone pain
* History of elevated CK
* Unexplained cramps
* Known sickle cell trait
* Cancer within the 5 years prior to study entry
* Diabetes
* Stroke, coronary artery or peripheral vascular disease
* Physical disability or previous injury interfering with exercise testing
* Pregnant or breastfeeding
* Depression (in last 3 years) or treatment with antidepressants
* Use of anti-psychotic drugs
* Alcohol abuse

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in pain score | Change from baseline at 2 months
Change in muscle function testing | Change from baseline at 2 months
  Strenght and endurance evaluation

SECONDARY OUTCOMES:
Change in muscle histology | Change from baseline at 2 months
  Histological, ultrastructural and metabolic assessment of muscle biopsy.
Change in pain score | Change from baseline at 5 months
Change in muscle function testing | Change from baseline at 5 months
Change in muscle histology | Change from baseline at 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Denis R Joanisse, PhD, Principal Investigator — Laval University; Jean Bergeron, MD, Principal Investigator — CHU de Quebec-Universite Laval; Jérôme Frenette, PhD, Principal Investigator — CHU de Quebec-Universite Laval
Locations (1):
- Centre hospitalier universitaire de Québec - CHUL, Québec, Quebec, Canada

REFERENCES:
- [Derived] Peyrel P, Mauriege P, Frenette J, Laflamme N, Greffard K, Dufresne SS, Huth C, Bergeron J, Joanisse DR. Impact of statin withdrawal on perceived and objective muscle function. PLoS One. 2023 Jun 14;18(6):e0281178. doi: 10.1371/journal.pone.0281178. eCollection 2023. PMID 37315062